CLINICAL TRIAL: NCT06303401
Title: Comparison of Thrust Manipulation of Sacroiliac Joint and Pelvic Stabilization Exercises on Pain and Disability Among Patients With Post-Partum Low Back Pain.
Brief Title: Comparison of Thrust Manipulation of Sacroiliac Joint and Pelvic Stabilization Exercises in Post Partum Low Back Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/MS-PT/01787 Gullalay
Record Dates: First submitted 2024-03-04; First posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Low Back Pain, Post Partum
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SI joint thrust Manipulation (Experimental): The patient was supine and the therapist stood contralateral to the side which was to be manipulated. The patient was passively moved into side bending toward the side to be manipulated. The therapist passively rotated the patient, and then delivered a quick thrust to the Anterior Superior Iliac Spine (ASIS) in a posterior and inferior direction
  Interventions: Other: SI joint thrust manipulation
- Pelvic Stabilization Exercises (Active Comparator): Heating pad for 10- 15 mints Pelvic stabilization exercises. Bridging (3 sets x 10 reps with 10 secs hold), Pelvic Tilt exercise (3 sets x 10 reps with 10 secs hold), Bird-Dog Exercise (3 sets x 10 reps with 10 secs hold), clamshell Exercise (3 sets x 10 reps with 10 secs hold).
  Interventions: Other: pelvic stabilization exercises

INTERVENTIONS:
Other: SI joint thrust manipulation — experimental group given the thrust manipulation along with heating pad. 3 sessions per week will be given for 4 weeks. The pain measure by using NPRS, functional status and disability through ODI will be evaluated.
  after every 3 sessions.
  Arms: SI joint thrust Manipulation
Other: pelvic stabilization exercises — Heating pad for 10- 15 mints Pelvic stabilization exercises include Bridging (3 sets x 10 reps with 10 secs hold) Pelvic Tilt exercise(3 sets x 10 reps with 10 secs hold) Bird-Dog Exercise (3 sets x 10 reps with 10 secs hold) clamshell Exercise (3 sets x 10 reps with 10 secs hold) .3 sessions per week will be given for 4 weeks. The pain using NPRS , functional status and disability will be evaluated by using ODI after every 3 sessions.
  Arms: Pelvic Stabilization Exercises

SUMMARY:
compare the effectiveness of SI joint thrust manipulation and pelvic stabilization exercises on Modified OSWESTRY Low Back pain Index (ODI) and Numeric Pain Rating Scale (NPRS) in patients with post-partum lower back pain.

DETAILED DESCRIPTION:
Patients fulfilling the inclusion criteria will be divided into 2 groups i.e. Group A and Group B. Patients in Group A will receive thrust manipulation technique and Group B will receive pelvic stabilization exercises, heating pad will be given to both groups. Patients will be treated 3 times per week for 4 consecutive weeks. Patient will be evaluated at baseline, midline and at end of 4th week. Pain, functional status and disability will be evaluated after every 3 sessions.

ELIGIBILITY:
Inclusion Criteria:

* age 20-40 years
* Postpartum women (after 6 weeks)(3, 12)
* Postpartum LBP patient
* Patient pain increased by provocation test i.e. Faber test, High thrust test and Gaenslen test

Exclusion Criteria:

* C-section
* inflammatory or malignant type of pain
* Neurological deficit
* Severe trauma
* Pelvic fracture
* Osteoporosis, spinal stenosis, spondylolysis, spondoloesthesisi

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Estimated)
Dates: Start 2023-09-27 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-08-30 (Estimated)

PRIMARY OUTCOMES:
Numeric pain rating scale (NPRS) | 4th week
  The Numeric Pain Rating Scale (NPRS) measures the subjective intensity of pain. The NPRS is an eleven-point scale: the patient rates pain from 0 (no pain) to 10 (worst imaginable pain).
Modified Oswestry Disability Index (ODI) | 4th week
  The ODI is a disease specific disability measure is used to establish a level of disability stage on a patient activity status and monitor change over the time. The ODI is made up of 10 questions. Each question is scored from (o-5) minimum to maximum.

CONTACTS AND LOCATIONS:
Overall Officials: Asmar Fatima, MS OMPT, Principal Investigator — Riphah International University
Locations (1):
- Lady Reading Hospital and Shahab Orthopedic & General Hospital, Peshawar, KPK, Pakistan

IPD SHARING:
Plan to Share IPD: No